CLINICAL TRIAL: NCT04369599
Title: Trans Thoracic Manipulation of Ventilation/Perfusion: the V/Q System
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: Georgia Tech Research Foundation (Unknown); Georgia Clinical & Translational Science Alliance (Unknown)
Responsible Party: Principal Investigator, Maxwell Weinmann, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: STUDY00000402
Record Dates: First submitted 2020-04-28; First posted 2020-04-30 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-05

CONDITIONS: Acute Respiratory Distress Syndrome; COVID-19
MeSH Terms: conditions — Respiratory Distress Syndrome; COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- V/Q System (Experimental): Participants with acute respiratory failure will undergo therapy with the V/Q System.
  Interventions: Device: V/Q System

INTERVENTIONS:
Device: V/Q System — With the patient supine, sedated, and hemodynamically stable, the Vest is placed upon the patient and secured by clinicians and staff. All chambers of the Vest will be inflated simultaneously. First inflation will be for one hour to a pressure of 0.4 psi. Subsequent inflations at 0.8 and finally 1.2 psi will be performed for one hour each. Participants will be treated for up to four hours and then will be observed for an additional hour.

SUMMARY:
The purpose of this pilot study is to measure the impact of non-invasive pneumatic manipulation of transthoracic pressure on oxygenation in patients with Acute Respiratory Distress Syndrome (ARDS) due to Coronavirus Disease 2019 (COVID 19) who are on mechanical ventilator support. This will be achieved by a pneumatic Vest placed around the chest wall of consenting patients who meet inclusion criteria. The Vest is essentially a non-invasive segmental device placed upon the anterior and posterior right and left aspects of the chest wall. The researchers have the ability to inflate and deflate the chambers of the Vest to achieve preset pressures as determined by the protocol and observe the patient's physiological response. Participants will have up to four hours of intervention with the study intervention, followed by 1 hour of post-intervention observation.

DETAILED DESCRIPTION:
Since the severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) surfaced at the end of 2019, transmission has been rapid and particularly lethal. Death is most commonly due to ARDS which has been quoted as occurring in up to 42% of patients. The rapid lethality of the COVID-19 has emphasized the limitations of currently available therapies in the Intensive Care Unit. Traditional mechanical ventilator support, the use of inhaled and systemic pulmonary vasodilatory drugs, invasive monitoring, proning and extracorporeal membrane oxygenation (ECMO) to name a few, are all voracious consumers of resources and have culminated in at least $27 billion expenditure per annum in the US alone pre-virus. This fiscal burden has been far exceeded in the current pandemic. With patient numbers growing exponentially hospital resources are being rapidly surpassed with ICU's overflowing which is exacerbated by a national shortage of mechanical ventilators. New techniques are demanded to both treat patients and identify responders if medical resources are to be optimized.

Traditionally, patients present to the ICU and are intubated once a threshold of respiratory distress and failure is reached. Various maneuvers are initiated to optimize oxygen uptake by the lungs to prevent the onset of organ failure and death. At present, there are no effective bridging technologies providing intervention between intubation to these costly more complex techniques which are almost solely the purview of more technologically adept tertiary academic centers. Clinical practice is often empiric and driven by trial and error in this emerging disease, largely because there are presently no clinical tests to provide clinicians with any clear indication as to which and whether patients will respond to these more costly difficult procedures. This is in part due to the underlying pathophysiology of ARDS where there is a further "uncoupling" between bloodflow,(and hence uptake of oxygen), and healthy lung units which allow transfer and absorption of oxygen because of the damage to the alveoli. This phenomenon shifts physiologic Ventilation/Perfusion mismatch (V/Q mismatch) into a pathologic state. Since this phenomenon is worsened by diseased tissue, it is diffuse but, not uniform and response to therapy is difficult to determine based on current modalities. Thus, many therapies are therefore instituted purely by trial and error. Determination of appropriate candidates for advanced therapeutic techniques is critically important as they are not without risk and resource consumption. Patients who are profoundly hypoxic and fail traditional supine position support are "flipped" onto their abdomen to assume the prone position, a technique known as proning. This requires a team of at least 6 nurses, respiratory therapists and physicians who attempt to ensure that there are no adverse events. Such complications contribute to the morbidity and potential mortality of the maneuver and include accidental extubation (displacement of the endotracheal tube out of the trachea), disconnection from the ventilator, transient worsening hypoxia, hemodynamic instability, dislodgement of central and peripheral venous catheters to name a few. This is further compounded by the need for greater sedation which is itself associated with hemodynamic instability, aspiration, altered conscious state and an increase in acuity of monitoring making it much more labor intensive and expensive.

The researchers propose the development of a ventilation/ perfusion system, (V/Q System), a pneumatically driven device which can improve oxygenation by adjusting trans-thoracic pressure gradients. This is a new field of lung physiology which is only just being explored. However, the concept of noninvasive manipulation of lung mechanics and ventilation/perfusion mismatch is profoundly impactful as it potentially introduces a comparatively safe technique to address an otherwise fatal failure of lung function. The V/Q System represents an effort to optimize lung function without the risk of patient proning. If successful, improved oxygenation associated with the device has multiple clinical and economic ramifications. Initially, the device may obviate the need to more costly, time consuming and potentially morbid procedures. Future research may include investigating if the device may be utilized to identify both "responders" and "non-responders" to advanced therapeutic techniques and can help eliminate the "trial and error" approach in managing complex ARDS patients.

The study procedures will take up to 5 hours to complete for each participant enrolled. During this time, the participant will be sedated per standard ICU protocol. Each study participant will have up to 4 hours of intervention with the study V/Q System, followed by 1 hour of post-intervention observation.

ELIGIBILITY:
Inclusion Criteria:

* Presentation with acute respiratory distress syndrome (ARDS) requiring intubation with mechanical ventilator support. ARDS will be defined by the ratio of the partial pressure of oxygen in the patient's arterial blood (PaO2) to the fraction of oxygen in the inspired air (FiO2) as being < 300.
* Ability of a Legally Authorized Representative (LAR) to provide consent on behalf of the patient.

Exclusion Criteria:

* Presence of cutaneous wounds that would be compromised by the Vest including stage 3 or greater pressure ulcers and the presence of actively treated burns
* Patients with pre-existing pulmonary hypertension and pulmonary fibrosis
* Bony chest trauma within the last 10 days
* Contraindications to esophageal manometry including recent esophageal trauma or surgery
* Abdominal compartment syndrome
* Active or recent gross hemoptysis
* Elevated intracranial pressure >20 mmHg
* LAR refusal to participate
* Severe Scoliosis
* Morbidly obese (BMI >37)
* Pregnant women
* Unable to maintain oxygen saturation > 88%

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2020-08-11 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Change in Arterial Oxygenation Levels | Baseline, Hour 1, Hour 2, Hour 3, Hour 4, 1 Hour Post-intervention
  Improvement in oxygenation will be assessed by a demonstrated >20% increase in arterial oxygen levels after 180 minutes of treatment with the V/Q Vest, with two different levels of pressure. Normal levels of arterial oxygen range from 75 to 100 millimeters of mercury (mm Hg). Low oxygenation levels necessitate supplemental oxygen.

CONTACTS AND LOCATIONS:
Overall Officials: Maxwell Weinmann, MD, Principal Investigator — Emory University
Locations (1):
- Emory University Hospital, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial will be made available for sharing, after deidentification.
Supporting Information: Study Protocol
Time Frame: Sharing of data will begin 9 months and end 36 months following article publication.
Access Criteria: Data will be made available for sharing with researchers who provide a methodologically sound proposal, in order to achieve aims stated in the approved proposal. Proposals may be submitted up to 36 months following article publication. After 36 months the data will be available in our University's data warehouse but without investigator support other than deposited metadata. Information regarding submitting proposals and accessing data may be found at (link to be provided).